CLINICAL TRIAL: NCT02808065
Title: Validation of Population Pharmacokinetic Model Derived From Healthy Volunteer in Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Yon Su Kim, Principal Investigator, Seoul National University Hospital
Other Study IDs: 17-2016-001-5
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplant; Kidney transplantation; Renal transplant; Renal transplantation
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tacrolimus + Mycophenolate mofetil
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Tacrolimus — Administered dose were individualized according to their own prescription
  Other Names: Prograf
Drug: Mycophenolate mofetil — Administered dose were individualized according to their own prescription
  Other Names: Cellcept

SUMMARY:
Pharmacokinetic model to predict interaction between tacrolimus and mycophenolate was developed through clinical trial with healthy volunteer. The purpose of this study is to confirm predictability of developed pharmacokinetic model in kidney transplant recipients.

DETAILED DESCRIPTION:
Study participants take their immunosuppressant as usual. One day, blood is drawn at predose and 1, 2, 3, 4-hour postdose to compare observed concentration with model-predicted concentration of tacrolimus and mycophenolate.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* At least 6 months after kidney transplantation
* Were on tacrolimus alone or tacrolimus plus mycophenolate based immunosuppressive regimen
* Maintained stable dose of immunosuppressants for at least two weeks

Exclusion Criteria:

* AST or ALT >3 upper limit of normal range
* Had gastrointestinal disorder that may affect an absorption of drug
* Coadministration of drugs that may affect the pharmacokinetics of immunosuppressive drug
* Multi-organ transplant recipient
* Severe psychiatric disorder
* Drug or alcohol abuser
* Pregnant
* Low compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus concentration | 0, 1, 2, 3, 4 hours post-dose

SECONDARY OUTCOMES:
Mycophenolate concentration | 0, 1, 2, 3, 4 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea